CLINICAL TRIAL: NCT00418847
Title: Pharmacokinetics and Tolerability of Zavesca® (Miglustat) In Patients With Juvenile GM2 Gangliosidosis: Single and Multiple Oral Doses
Brief Title: Pharmacokinetics and Tolerability of Zavesca® (Miglustat) In Patients With Juvenile GM2 Gangliosidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000004763
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Gangliosidoses GM2
Keywords: pediatrics; lysosomal storage diseases; Gangliosidoses GM2; Tay-Sachs disease; Sandhoff disease; Infantile GM2-activator deficiency; Miglustat
MeSH Terms: conditions — Gangliosidoses, GM2; Lysosomal Storage Diseases; Tay-Sachs Disease; Sandhoff Disease | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: miglustat

INTERVENTIONS:
Drug: miglustat — Target dose of 320 mg/m^2/day (divided in 3 doses) will be based on the Body Surface Area (BSA). For children with a BSA > 1.3, 200 mg TID will be administered. For children with a BSA of 0.8-1.3, 100 mg TID will be administered.
  Other Names: Zavesca

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics of Zavesca (miglustat, OGT918) when given as single and multiple doses in juvenile patients with GM2 gangliosidosis.

DETAILED DESCRIPTION:
The GM2 gangliosidoses are a group of neuro-degenerative lysosomal storage diseases resulting from accumulation of GM2 and related glycolipids in the central nervous system (CNS). Tay-Sachs and Sandhoff disease are two variants which are indistinguishable in clinical grounds. According to the onset and rate of disease progression, the condition can be categorized in infantile, juvenile and adult forms. This open-label, single-arm study is designed to assess the pharmacokinetics, safety and tolerability of miglustat in juvenile patients. Miglustat will be administered at a maximum dose of 600 mg/day, divided into three doses per day. The dose used for patients in this pediatric age range will be related to the patient's body surface area. The pharmacokinetics assessments for the study will be performed in-hospital during a 24 hour period, and will take place at the day one and at the month 3 visits. The clinical (which includes safety and tolerability) assessments will be performed throughout the 24-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GM2 gangliosidosis confirmed by demonstration of profound deficiency of β-hexosaminidase A or A & B in peripheral blood leukocytes or cultured skin fibroblasts
* Aged 6 to 20 years
* Onset of characteristic clinical symptoms of the disease before age 15 years
* Normal renal or hepatic function

Exclusion Criteria:

* Fertile patients who do not agree to use adequate contraception throughout the study and for 3 months after cessation of miglustat treatment.
* Patients who cannot tolerate the study procedures, cannot be compliant to therapy or who are unable to travel to the study center as required by this protocol.
* Patients receiving other investigational agents within 3 months of study initiation.
* Patients with disease that may affect absorption or elimination of drugs.
* Patients suffering from clinically significant diarrhea (>3 liquid stools per day for > 7 days) without definable cause within 3 months of baseline visit, or who have a history of significant gastrointestinal disorders.
* Patients with swallowing difficulties.
* Patients with a high probability of dying during the study.
* Patients who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2004-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Concentration of miglustat in plasma | Periodic intervals up to 24 hours

SECONDARY OUTCOMES:
Changes in volume loss and signal intensity from baseline MRI | 12 months
Change in single-voxel N acetylaspartate (NAA) from baseline MRS | 1 month, 3 months, 6 months, 9 months, and 12 months
Change in neuropsychological testing from baseline | 6 months and 12 months
Change in nerve conduction | 6 months and 12 months
Change in neurological examination from baseline | 1 month, 3 months, 6 months, 9 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joe TR Clarke, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Maegawa GH, Banwell BL, Blaser S, Sorge G, Toplak M, Ackerley C, Hawkins C, Hayes J, Clarke JT. Substrate reduction therapy in juvenile GM2 gangliosidosis. Mol Genet Metab. 2009 Sep-Oct;98(1-2):215-24. doi: 10.1016/j.ymgme.2009.06.005. Epub 2009 Jun 12. PMID 19595619